CLINICAL TRIAL: NCT03963713
Title: Stereotactic Radiotherapy and Conventionally-fractionated-image-guided Intensity Modulated Radiotherapy for Spinal Metastatic Tumors：A Prospective Multicenter Cohort Study
Brief Title: Stereotactic Radiotherapy and Image-guided Intensity Modulated Radiotherapy for Spinal Metastatic Tumors
Acronym: SCIRSM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Mianyang Central Hospital (Other); Second Hospital of Shanxi Medical University (Other); Qingdao chengyang hospital (Unknown); Qingdao Hiser Medical Group (Other); Beijing 302 Hospital (Other); Guangxi Ruikang Hospital (Other); Third Affiliated Hospital of Guizhou Medical University (Unknown); Panjin Liaohe Oilfield Gem Flower Hospital (Other); Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BYSY-CKIMRT-SPNALM
Record Dates: First submitted 2019-05-21; First posted 2019-05-28 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-05

CONDITIONS: Radiotherapy; Spine Metastases; Radiosurgery
Keywords: Stereotactic radiotherapy; Intensity modulated radiotherapy; spinal metastatic tumors
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: non-randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Stereotactic radiotherapy (Experimental): In this study, the metastases were treated with Stereotactic radiotherapy（SBRT）.Using multimodal image fusion to outline the target area.PTV = GTV + 0-10mm Target volume radiation dose: The range of BED value of radiotherapy was 60-72 when the distance between the tumor and gastrointestinal tract or spinal cord was more than 5 mm (alpha/beta=10) and 51.3-59.5 when the distance between the tumor and gastrointestinal tract or spinal cord was less than 5 mm (alpha/beta=10).
  Stereotactic radiotherapy
  Interventions: Radiation: Stereotactic radiotherapy
- Conventionally-fractionated image- guided Intensity modulated (Experimental): In this study, the metastases were treated with Conventionally-fractionated image- guided Intensity modulated radiotherapy.Using multimodal image fusion to outline the target area.The dose of the target volume radiotherapy dose is 30 Gy/10f or 40Gy/20f.Previous treatment and follow-up data will be analyzed to evaluate the clinical efficacy comparison of stereotactic radiotherapy and conventionally-fractionated image-guided intensity-modulated radiotherapy for spinal metastatic tumors, local control rate and side effects, and to clarify the effectiveness and safety of different doses of radiotherapy.
  Interventions: Radiation: Conventionally-fractionated image- guided Intensity modulated radiotherapy

INTERVENTIONS:
Radiation: Stereotactic radiotherapy — Using multimodal image fusion to outline the target area.PTV = GTV + 0-10mm Target volume radiation dose: The range of BED value of radiotherapy was 60-72 when the distance between the tumor and gastrointestinal tract or spinal cord was more than 5 mm (alpha/beta=10) and 51.3-59.5 when the distance between the tumor and gastrointestinal tract or spinal cord was less than 5 mm (alpha/beta=10).
  Arms: Stereotactic radiotherapy
Radiation: Conventionally-fractionated image- guided Intensity modulated radiotherapy — Using multimodal image fusion to outline the target area.The dose of the target volume radiotherapy dose is 30 Gy/10f or 40Gy/20f.Previous treatment and follow-up data will be analyzed to evaluate the clinical efficacy comparison of stereotactic radiotherapy and conventionally-fractionated image-guided intensity-modulated radiotherapy for spinal metastatic tumors, local control rate and side effects, and to clarify the effectiveness and safety of different doses of radiotherapy.
  Arms: Conventionally-fractionated image- guided Intensity modulated

SUMMARY:
Data of 100 patients with spinal metastatic tumor who received stereotactic radiotherapy or conventionally-fractionated image-guided intensity-modulated radiotherapy in the multi-center of the research group from July 2019 to June 2021 will be collected, as well as their follow-up data.Previous treatment and follow-up data will be analyzed to evaluate the clinical efficacy comparison of stereotactic radiotherapy and conventionally-fractionated image-guided intensity-modulated radiotherapy for spinal metastatic tumors, local control rate and side effects, and to clarify the effectiveness and safety of different doses of radiotherapy.

DETAILED DESCRIPTION:
In this study, Data of 100 patients with spinal metastatic tumor who received stereotactic radiotherapy or conventionally-fractionated image-guided intensity-modulated radiotherapy in the multi-center of the research group from July 2019 to June 2021 will be collected, as well as their follow-up data.The metastases were treated with SBRT.Using multimodal image fusion to outline the target area.PTV = GTV + 0-10mm Target volume radiation dose: The range of BED value of radiotherapy was 60-72 when the distance between the tumor and gastrointestinal tract or spinal cord was more than 5 mm (alpha/beta=10) and 51.3-59.5 when the distance between the tumor and gastrointestinal tract or spinal cord was less than 5 mm (alpha/beta=10).The metastases were treated with Conventionally-fractionated image- guided Intensity modulated radiotherapy.Using multimodal image fusion to outline the target area.The dose of the target volume radiotherapy dose is 30 Gy/10f or 40Gy/20f.Previous treatment and follow-up data will be analyzed to evaluate the clinical efficacy comparison of stereotactic radiotherapy and conventionally-fractionated image-guided intensity-modulated radiotherapy for spinal metastatic tumors, local control rate and side effects, and to clarify the effectiveness and safety of different doses of radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old;
* Spine metastatic tumor patients confirmed by pathology and imaging; Number 3; Surgical treatment is not possible due to iatrogenic or (and) personal factors;
* Spinal metastasis after previous systemic treatment or progression after previous treatment of spinal metastasis;
* The anatomy of the spinal metastases form Tomita parting Ⅰ type - Ⅲ type; Without systemic metastasis or metastasis, the lesion was controlled.
* ECOG physical condition score: 0-1, Karnofsky score 60, able to withstand puncture;
* Expected survival 3 months;
* Main organ function is good, without serious hypertension, diabetes and heart disease.
* Has signed informed consent;
* The compliance was good and the family members agreed to follow up for survival.

Exclusion Criteria:

* Of the anatomy of the spinal metastases form Tomita classification: Ⅳ, Ⅴ Ⅵ, Ⅶ.
* Participated in other drug clinical trials within four weeks; There was a history of bleeding, and any bleeding event with severe grade of CTCAE5.0 or above occurred within 4 weeks before screening;
* Screening of patients with known central nervous system metastasis or a history of central nervous system metastasis. For patients with clinical suspected central nervous system metastasis, CT or MRI examination must be performed within 14 days before randomization to exclude central nervous system metastasis.
* Patients with hypertension who cannot obtain good control by single antihypertensive drug treatment (systolic blood pressure >140mmHg, diastolic blood pressure >90mmHg); Having a history of unstable angina pectoris; Patients newly diagnosed with angina within 3 months before screening or myocardial infarction within 6 months before screening; Arrhythmia (including QTcF: 450ms in male and 470ms in female) requires long-term use of anti-arrhythmia drugs and New York heart association grade II cardiac dysfunction;
* Long-term unhealed wounds or incomplete fracture healing;
* Imaging showed that the tumor had invaded important blood vessels or the researchers judged that the patient's tumor had a very high possibility to invade important blood vessels during the treatment and cause fatal bleeding;
* Coagulation function is unusual, have haemorrhage tendency person (before random 14 days must satisfy: below the circumstance that does not use anticoagulant INR is in normal value range); Patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or their analogues; The use of low-dose warfarin (1mg oral, once daily) or low-dose aspirin (no more than 100mg daily) for preventive purposes is permitted on the premise that the international standardized ratio of prothrombin time (INR) is 1.5;
* Screening for the occurrence of hyperactive/venous thrombosis events in the first 6 months, such as cerebrovascular accidents (including temporary ischemic attack), deep vein thrombosis (except for venous thrombosis caused by intravenous catheterization in the early stage of chemotherapy, which was determined by the researchers to have recovered) and pulmonary embolism, etc.
* Thyroid function was abnormal in the past and could not be kept within the normal range even in the case of drug treatment.

  (10) Attending has a history of psychotropic drug abuse, and can't attend or has mental disorder;
* Always half a year after spinal tumors or other close to the spine tumor lesion lesions radiation;
* Immunodeficiency disease, or has other acquired, congenital immunodeficiency disease, or has a history of organ transplantation;
* Judgment according to the researchers, there is serious to endanger the safety of patients or patients completed the research associated with disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-06-10 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Cancer pain score | 1 year after the treatment
  Numerical grading (NRS) should be used for pain intensity assessment, and facial expression pain scoring should be used for patients with difficulty in expression.
Muscle strength and muscle tension grading | 1 year after the treatment
  Muscle strength and muscle tension were graded by Numbers
JOA score of cervical and lumbar vertebrae | 2 years after the treatment
  JOA score of cervical and lumbar vertebrae
Quality of Life Score of Tumor Patients(0-60) | 2 years after the treatment
  Common methods for evaluating the quality of life of patients:The full score of quality of life is 60, the worst is < 20, the worse is 21-30, the average is 31-40, the better is 41-50, and the good is 51-60.

SECONDARY OUTCOMES:
Duration of pain response | 1 years after the treatment
  Time from complete or partial pain relief to pain worsening (≥ 3 points on the NRPS
Overall survival | 3 years after the treatment
  The time from enrollment to death from any cause
Local control rate | 3 years after the treatment
  The rate at which lesions remained stable during follow-up
Adverse reactions | 6 months after the treatment
  Adverse reactions during and after treatment
Progression-free survival | 3 years after the treatment
  Time from treatment to cancer progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Junjie Wang, MD, Study Chair — Peking University Third Hospital; Fei Xu, M Med, Study Director — Peking University Third Hospital; Hongqing Zhuang, M Med, Principal Investigator — Peking University Third Hospital; Xiaobo Du, MD, Principal Investigator — Mianyang Central Hospital; Jie Li, M Med, Principal Investigator — Mianyang Central Hospital; Xiang Song, M Med, Principal Investigator — Second Hospital of Shanxi Medical University; Lei Zhang, M Med, Principal Investigator — Second Hospital of Shanxi Medical University; Jianguo Zhang, M Med, Principal Investigator — Qingdao chengyang people's hospital; Peng Liu, M Med, Principal Investigator — Qingdao Hiser Medical Group; Xuezhang Duan, MD, Principal Investigator — Beijing 302 Hospital; Zuping Lian, MD, Principal Investigator — Guangxi Ruikang Hospital; Liang Liu, MD, Principal Investigator — Third Affiliated Hospital of Guizhou Medical University; Longhai Shen, M Med, Principal Investigator — Panjin Liaohe Oilfield Gem Flower Hospital; Dongjie He, M Med, Principal Investigator — Tang-Du Hospital; Xuemin Li, MD, Principal Investigator — Peking University Third Hospital; Yi Chen, MD, Principal Investigator — Peking University Third Hospital
Locations (10):
- China (10):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The fifth medical center of PLA general hospital, Beijing, Beijing Municipality
  - Guangxi ruikang hospital, Nanning, Guangxi
  - Third Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - GEM flower hospital of Liaohe oil field Tang-Du Hospital, Panjin, Liaoning
  - Hiser Medical Center of Qingdao, Qingdao, Shandong
  - Qingdao chengyang people's hospital, Qingdao, Shandong
  - Second hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Tangdu hospital, Xian, Shanxi
  - Mianyang Central Hospital, Mianyang, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Massicotte E, Foote M, Reddy R, Sahgal A. Minimal access spine surgery (MASS) for decompression and stabilization performed as an out-patient procedure for metastatic spinal tumours followed by spine stereotactic body radiotherapy (SBRT): first report of technique and preliminary outcomes. Technol Cancer Res Treat. 2012 Feb;11(1):15-25. doi: 10.7785/tcrt.2012.500230. PMID 22181327
- [Background] Sahgal A, Whyne CM, Ma L, Larson DA, Fehlings MG. Vertebral compression fracture after stereotactic body radiotherapy for spinal metastases. Lancet Oncol. 2013 Jul;14(8):e310-20. doi: 10.1016/S1470-2045(13)70101-3. PMID 23816297
- [Background] Rades D, Stalpers LJ, Veninga T, Schulte R, Hoskin PJ, Obralic N, Bajrovic A, Rudat V, Schwarz R, Hulshof MC, Poortmans P, Schild SE. Evaluation of five radiation schedules and prognostic factors for metastatic spinal cord compression. J Clin Oncol. 2005 May 20;23(15):3366-75. doi: 10.1200/JCO.2005.04.754. PMID 15908648
- [Background] Gong Y, Wang J, Bai S, Jiang X, Xu F. Conventionally-fractionated image-guided intensity modulated radiotherapy (IG-IMRT): a safe and effective treatment for cancer spinal metastasis. Radiat Oncol. 2008 Apr 22;3:11. doi: 10.1186/1748-717X-3-11. PMID 18426607
- [Background] Guckenberger M, Goebel J, Wilbert J, Baier K, Richter A, Sweeney RA, Bratengeier K, Flentje M. Clinical outcome of dose-escalated image-guided radiotherapy for spinal metastases. Int J Radiat Oncol Biol Phys. 2009 Nov 1;75(3):828-35. doi: 10.1016/j.ijrobp.2008.11.017. Epub 2009 Feb 26. PMID 19250762
- [Background] Zhang M, Chen YR, Chang SD, Veeravagu A. CyberKnife stereotactic radiosurgery for the treatment of symptomatic vertebral hemangiomas: a single-institution experience. Neurosurg Focus. 2017 Jan;42(1):E13. doi: 10.3171/2016.9.FOCUS16372. PMID 28041316
- [Background] Gandhidasan S, Ball D, Kron T, Bressel M, Shaw M, Chu J, Chander S, Wheeler G, Plumridge N, Chesson B, David S, Siva S. Single Fraction Stereotactic Ablative Body Radiotherapy for Oligometastasis: Outcomes from 132 Consecutive Patients. Clin Oncol (R Coll Radiol). 2018 Mar;30(3):178-184. doi: 10.1016/j.clon.2017.11.010. Epub 2017 Dec 8. PMID 29224900
- [Background] Ryu S, Rock J, Rosenblum M, Kim JH. Patterns of failure after single-dose radiosurgery for spinal metastasis. J Neurosurg. 2004 Nov;101 Suppl 3:402-5. PMID 15537196
- [Background] Chang EL, Shiu AS, Mendel E, Mathews LA, Mahajan A, Allen PK, Weinberg JS, Brown BW, Wang XS, Woo SY, Cleeland C, Maor MH, Rhines LD. Phase I/II study of stereotactic body radiotherapy for spinal metastasis and its pattern of failure. J Neurosurg Spine. 2007 Aug;7(2):151-60. doi: 10.3171/SPI-07/08/151. PMID 17688054
- [Background] Gerszten PC, Burton SA, Ozhasoglu C, Welch WC. Radiosurgery for spinal metastases: clinical experience in 500 cases from a single institution. Spine (Phila Pa 1976). 2007 Jan 15;32(2):193-9. doi: 10.1097/01.brs.0000251863.76595.a2. PMID 17224814
- [Background] Wowra B, Zausinger S, Drexler C, Kufeld M, Muacevic A, Staehler M, Tonn JC. CyberKnife radiosurgery for malignant spinal tumors: characterization of well-suited patients. Spine (Phila Pa 1976). 2008 Dec 15;33(26):2929-34. doi: 10.1097/BRS.0b013e31818c680a. PMID 19092627
- [Background] Expert Panel on Radiation Oncology-Bone Metastases; Lo SS, Lutz ST, Chang EL, Galanopoulos N, Howell DD, Kim EY, Konski AA, Pandit-Taskar ND, Rose PS, Ryu S, Silverman LN, Sloan AE, Van Poznak C. ACR Appropriateness Criteria (R) spinal bone metastases. J Palliat Med. 2013 Jan;16(1):9-19. doi: 10.1089/jpm.2012.0376. Epub 2012 Nov 20. PMID 23167547